CLINICAL TRIAL: NCT06920797
Title: Evaluation of New Strategies in the Analysis of the Reproductive Tract Microbiome: A Descriptive Pilot Study
Brief Title: New Strategies to Evaluate the Reproductive Tract Microbiome
Acronym: niMICROBIOME
Status: Recruiting | Type: Observational
Sponsor: Igenomix (Industry)
Responsible Party: Sponsor
Other Study IDs: IGX1-MIC-DV-24-04
Record Dates: First submitted 2025-03-17; First posted 2025-04-10 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Fertility; Infertility; Reproductive Health; Microbiome Analysis
Keywords: endometrial microbiome; Microbiome; Reproductive tract; Pathogenic bacteria; Dysbiosis
MeSH Terms: conditions — Infertility; Dysbiosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Endometrial and vaginal microbiome description: Participants in this group will undergo two rounds of samples collection, 1, 2 or 3 months apart, as assigned by the investigator.
  Interventions: Diagnostic Test: Reproductive tract microbiome analysis

INTERVENTIONS:
Diagnostic Test: Reproductive tract microbiome analysis — Assessment of the endometrial and vaginal microbiome in three different samples: endometrial biopsy (EB), endometrial fluid (EF) and vaginal swab (VS).

SUMMARY:
The goal of this observational study is to evaluate alternative less invasive sampling methods for the analysis of the endometrial microbiome. For that, vaginal swab and endometrial fluid samples will be assessed in comparison with the standard sampling method (an endometrial biopsy), in women aged 18-50 years on an oocyte donation program and/or who attend the clinic for routine gynecological controls, and whose samples will be collected during the secretory phase of a natural menstrual cycle. The study aims to:

* Evaluate the pontential of the less invasive techniques to assess the endometrial microbiome, compared to the endometrial biopsy, as well as their safety.
* Evaluate the microbiome's stability in a period of 1 to 3 months.

Participants will undergo a sampling round (of the 3 sampling methods), and then a second round 1, 2 or 3 months later, as assigned by the investigator.

DETAILED DESCRIPTION:
The endometrium plays a pivotal role in reproductive health, influencing processes such as implantation and pregnancy. Although the endometrium has generally been considered a tissue free of bacteria, numerous studies have documented the presence of an endometrial microbiome mainly composed of different species from the Lactobacillus genus. The presence of pathogenic bacteria has been shown to disrupt the uterine environment, affecting implantation rates and pregnancy success.

Traditional and emerging sampling methods allow for the study of the microbial profile of the endometrium, but the efficiency and representativeness of these techniques vary. Therefore, this study aims to compare the effectiveness, accuracy, and usefulness of three different sampling methods for microbiome analysis: endometrial biopsy, endometrial fluid, and vaginal swab. Additionally, it seeks to compare the endometrial microbial profiles with the vaginal microbiome to assess whether it may provide indirect information about the upper reproductive tract.

Endometrial biopsy is a gynecological procedure routinely performed in the clinical practice to provide the patient with an analysis of their microbiome before embryo transfer, ensuring that it is carried out in a non-pathological endometrium, especially in patients with previous implantation failures. It is considered the standard for uterine lining sampling but is an invasive technique that, due to the discomfort associated with the procedure itself, may not always be feasible. Endometrial fluid is a less invasive method that offers a potential alternative by collecting cells from the endometrial surface. On the other hand, studying the vaginal microbiome, although it may provide insight into reproductive outcomes, may not accurately reflect the microbiome of the uterine cavity, a key location where implantation and pregnancy occur. By using comprehensive microbiome analysis techniques, this study will assess the microbial populations collected by each method and determine the efficiency and usefulness of each sampling technique.

Through direct comparison, this research aims to establish a clearer understanding of how sampling techniques can impact microbiome analysis in the context of reproductive health. The results obtained could have significant implications for clinical practice, potentially offering less invasive and more accurate methods to evaluate the endometrial microbiome. This study aims not only to redirect our approach to sampling the endometrial microbiome but also to improve our understanding of its role in female reproductive health. Furthermore, it would facilitate the assessment of potential correlations between the endometrial and vaginal microbiomes.

ELIGIBILITY:
Inclusion Criteria:

* Women, between 18 and 50 years, coming form the donor program and/or patients from the General Gynaecology Unit who attend to routine gynaecological controls to the clinic and who voluntarily accept to participate and sign the corresponding informed consent approved by the Ethics Committee, once they have been dully informed of the study's nature and knoe the potential risks, benefits and discomforts.

Exclusion Criteria:

* Ongoing pregnancy.
* Samples not obtained during the secretory phase of a natural cycle.
* Intake of any antibiotic, probiotic and/or antifungal in the 7 days prior to the sample collection of the first cycle.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women, between 18 and 50 years, coming form the donor program and/or patients from the General Gynaecology Unit who attend to routine gynaecological controls to the clinic, and whose samples will be taken during the secretory phase of the natural menstrual cycle.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-06-09 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Evaluation of minimally invasive techniques for the analysis of the endometrial microbiome | From enrollment to the second sampling round (1 to 3 months, depending on the study assigned group))
  Assessment of the viability and technical reliability of the new sampling techniques (endometrial fluid -EF- and vaginal swab -VS-) to evaluate the endometrial microbiome, compared with the standard sampling technique, the endometrial biopsy - EB-. The endometrial microbiome composition will be determined by DNA extraction and bacterial profiling from the three samples (endometrial biopsy -EB-, endometrial fluid -EF- and vaginal swab -VS-). The EB microbiome will serve as reference and it will be compared with the EF's and VS's microbiome to determine whether they are equivalent.

SECONDARY OUTCOMES:
Evaluation of the inter-cycle consistency of the microbial profile in a period of 1 to 3 months | From enrollment to the second sampling round (1 to 3 months, depending on the study assigned group))
  Comparison of the endometrial microbiome from each patient at 2 different time points, 1, 2 or 3 months apart. The endometrial microbiome of each patient, determined by DNA extraction and bacterial profiling of the three samples, will be compared at two different time points (1, 2 or 3 months apart) to determine the microbiome's and technique stability and robustness.
Safety evaluation of the sampling techniques (EB, EF and VS) | From enrollment to the end of the study (from 1 to 3 months, depending on the assigned group)
  Registration of any relevant adverse events related to the techniques reported by participants

OTHER OUTCOMES:
Correlation of the VS's and EF's pH with the microbiome | From enrollment to the second sampling round (1 to 3 months, depending on the study assigned group))
  Determination of the pH in the VS and EF samples and assessment of the possible correlation with the microbial profile.

CONTACTS AND LOCATIONS:
Locations (1):
- Vida Recoletas Sevilla, Seville, Seville, Spain

IPD SHARING:
Plan to Share IPD: No